CLINICAL TRIAL: NCT03051854
Title: Prevalence, Consequences and Prevention of Violence Against Children in Southwestern Uganda
Brief Title: Prevention of Violence Against Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Bielefeld University (Other); Alexander von Humboldt Association (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Elbert, Professor for Clinical Psychology and Behavioural Neuroscience, University of Konstanz
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ICC-T-2017-Uganda
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Violence Against Children
Keywords: Violence; Children; Prevalence; Abuse; Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICC-T (Experimental): Intervention: Interaction Competencies with children - for teachers (ICC-T) 5.5 days with 8 hours of training for teachers. Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Interventions: Behavioral: Interaction Competencies with children - for teachers
- Control schools (No Intervention): The control school do not receive any intervention.

INTERVENTIONS:
Behavioral: Interaction Competencies with children - for teachers — Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting.
  Arms: ICC-T

SUMMARY:
Beside the home, the school is often the second important setting for the development and education of children and adolescents. Students spend a large part of their life at school. However, there is recurrent occurrence of violence against children and of harsh discipline measures used in home and school settings. These may result into negative consequences. Hence, prevention strategies against the use of harsh discipline use in schools become a priority.

In the baseline of this study the investigators will therefore examine the prevalence and consequences of violence against children in Southwestern Uganda. The study will be conducted in schools and common disciplinary measures used by teachers, and the perceptions of teachers' and students' in relation to commonly used and experienced disciplinary measures we will be investigated.

In the second phase, the investigators then will implement and assess the effectiveness of an intervention aimed at reducing the use of harsh and violent disciplinary measures in schools. ICC-T training in the long-term aims at fostering better relations amongst students and teachers. Based on feasibility studies, ICC-T intervention is expected to result into better teacher-student relationships, change in teachers' attitudes and behaviors concerning the use of violent disciplinary measures in the school setting.

DETAILED DESCRIPTION:
Study participants (i.e., teachers and students) will be recruited from six districts in southwestern Uganda. The sample will include 12 government-aided secondary schools from which 60 students and 15-25 teachers will be recruited. The final sample will have 720 students and 180-300 teachers. Investigators will assess data in the baseline (i.e., prior to intervention) and three months after the intervention.

Study measures will cover the following topics: socio-demographic data, common disciplinary measure used at home and at school, students' mental health problems, students' and teachers' attitudes towards violent discipline measures, and students' exposure to peer and sexual violence. Questionnaire for teachers will have additional items that measure attitudes towards teaching and teacher stress. Additionally, the investigators will also assess the demand, acceptance and feasibility of the training.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (if underaged by parents & minors)

Exclusion Criteria:

* Acute drug or alcohol intoxication
* Acute psychotic disorder

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in teachers' application of harsh discipline | The CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  In teachers the Conflict Tactics Scale Parent-Child version (CTSPC) will assess teachers' use of violent discipline measure against students in the school locale.
Change in student's exposure to harsh discipline by teachers | CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Conflict Tactics Scale Parent-Child version (CTSPC) will assess the students' self-reported experiences of violent discipline in schools.

SECONDARY OUTCOMES:
Change in student's mental health | SDQ will be used at (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  Strength and Difficulties Questionnaire (SDQ) will assess students' internalizing and externalizing problems. SDQ will be used at T1 and T2.
Change in teachers's attitudes towards harsh discipline | The adapted version of CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  Items of the CTSPC have been adapted to measure teachers' and students' attitudes towards violent discipline methods at school.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hecker, PhD, Principal Investigator — Bielefeld University
Locations (1):
- Government-aided secondary schools, Mbarara, Southwestern Uganda, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ssenyonga J, Hermenau K, Nkuba M, Hecker T. Reducing violence against children by implementing the preventative intervention Interaction Competencies with Children for Teachers (ICC-T): study protocol for a cluster randomized controlled trial in Southwestern Uganda. Trials. 2018 Aug 13;19(1):435. doi: 10.1186/s13063-018-2827-9. PMID 30103776